CLINICAL TRIAL: NCT07391956
Title: TIER-PALLIATIVE CARE: A Population-based Care Delivery Model to Match Evolving Patient Needs and Palliative Care Services for Community-based Patients With Heart Failure or Cancer
Brief Title: Tier Palliative Care For Patients With Advanced Heart Failure or Cancer
Acronym: TIER-PC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Laura Gelfman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY-22-00591 R01
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Heart Failure; Advanced Non-Colorectal Gastrointestinal Cancer; Advanced Lung Cancer; Advanced Triple Negative Breast Cancer
Keywords: palliative care; community-based; advanced heart failure; advanced cancer
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tier-Palliative Care (Experimental): Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician based on symptom burden and function.
  Interventions: Behavioral: Tier-Palliative Care
- Augmented Control (Active Comparator): Visits to the patient from a CHW without training in heart failure, cancer or palliative care.
  Interventions: Behavioral: Community Health Worker

INTERVENTIONS:
Behavioral: Tier-Palliative Care — TIER-PC is an adaptive model of delivering palliative care that provides the right level of care to the right patients at the right time. TIER-PC increases the number and intensity of disciplines added to the patient's care team as their symptoms worsen and function declines.
  Other Names: Tier-PC
  Arms: Tier-Palliative Care
Behavioral: Community Health Worker — Usual Care plus the addition of a community health worker who will serve as a health coach for the participant.
  Arms: Augmented Control

SUMMARY:
TIER-PC is an adaptive model of delivering palliative care that provides the right level of care to the right patients at the right time. It represents an adaption of the Mount Sinai PALLIATIVE CARE AT HOME (PC@H) program, which delivers home-based palliative care. TIER-PC increases the number and intensity of disciplines added to the patient's care team as their symptoms worsen and function declines. In Tier 1, patients who are able to care for themselves and no/mild symptoms receive a community health worker (CHW) trained to elicit illness understanding in a culturally competent way. In Tier 2, for patients with poorer function and mild symptoms, a social worker (SW), trained in serious illness communication, joins the CHW to further elicit patients' goals and prognostic understanding while communicating symptom needs to their primary clinician. In Tier 3, as function decreases and symptoms increase, an advance practice nurse (APN) joins the CHW and SW to manage complex symptoms. Finally, in Tier 4, for those older adults with the poorest function and most complex symptoms, a physician joins the team to ensure that the most complex needs (e.g., end-of-life treatment preferences and multifaceted symptom control) are met. The CHW follows patients longitudinally across all tiers and re-allocates them to the appropriate tier based on their evolving needs.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to study the impact of a novel home based palliative care intervention on patients' symptoms, quality of life, and completion of goals of care documentation. In addition, the study will examine the impact of this model of care on patient healthcare utilization, including hospitalization, emergency department utilization, and hospice use prior to death. The trial will also include patients' caregivers, in order to examine the impact of the intervention on caregiver anxiety, satisfaction with care and post-traumatic symptoms. Patients randomized to the intervention will be scheduled for Tier-PC visit community health work to allocate to Tier-PC tier. Visits will combine a combination of video-teleconferencing technology and in person visits. Patients in the intervention arm will receive ongoing monitoring and input (telephone-based, video-based, and in-person) from members of the clinical team, dependent on their identified needs. Patients' cases will be discussed at the weekly IDT meeting, as appropriate to the level of clinical need. Patients and caregivers will be provided with access to a 24 hour telephone line, staffed by a Mount Sinai based physician, which acts as an advice line out of hours. These physicians will be able to provide advice to patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Heart Failure (HF) with two HF-related hospitalizations within the last 12 months or
* Advanced lung or non-colorectal gastrointestinal cancer (pancreatic, gastric, hepatobiliary, small bowel, esophageal) or tripe negative breast cancer with one hospitalization within the last 6 months
* KPS > or = 50% (ECOG 0, 1 or 2)
* > 2 outpatient MSHS visits in prior 12 months
* Manhattan or Queens residence
* Capacity to provide informed consent
* English or Spanish fluency
* > or = 18 years of age

Exclusion Criteria:

* Diagnoses of both cancer and advanced HF
* Lung cancer with a driver mutation (e.g., EGFR) that confers a favorable prognosis and does not follow typical trajectory
* Patients with > 1 visit to Outpatient Supportive Oncology/Cardiology visit
* Patients with last visit to Outpatient Supportive Oncology/Cardiology < 3 months ago
* Previous receipt of a ventricular assist device or previous heart transplantation
* Receiving hospice care prior to study enrollment or enrolled in another study of a palliative care patient/caregiver intervention
* Living in a facility (subacute rehab, long-term care facility, hospice facility or residence)
* Callahan 6-Item Cognitive Screening score ≤3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) | 12 months
  Patient symptoms: Edmonton Symptom Assessment Scale (ESAS), 9 items, each item is scored on a 10-point scale, total score ranges from 0-90, higher scores indicate more symptoms.
Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-Pal) | 12 months
  Patient quality of life: Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-Pal), a 46-item QoL questionnaire validated in patients with advanced disease. Each item is scored on a 5-point likert scale. Total score ranges from 0-184, higher scores indicate better quality of life
Patient-reported goals of care discussion | 12 months
  Patient-reported Goals of Care Discussions: "Have you ever discussed with this doctor the kind of medical care you would want if you were too sick to speak for yourself?" Response: Yes/No

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 12 months
  Generalized Anxiety Disorder-7 (GAD-7), a 7-item scale, Full scale from 0-21, higher scores indicates more anxiety.
Family Satisfaction with End-of-Life Care (FAMCARE-10) | 12 months
  FAMCARE-10 to assess caregiver satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. Full scale ranges 0-20, with higher scores indicating higher satisfaction.
Number of hospital admissions | 12 months
  Number of hospital admissions: Acute care utilization as measured by the number of hospital admissions
Number of hospital days | 12 months
  Number of hospital days: Acute care utilization as measured by the number of hospital days
Number of emergency department (ED) visits | 12 months
  Number of emergency department (ED) visits: Acute care utilization as measured by the number of ED visits

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gelfman, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Mount Sinai Queens, Astoria, New York
  - Mount Sinai Downtown, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Morningside, New York, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to Christian.Espino@mssm.edu
  . To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).